CLINICAL TRIAL: NCT06897137
Title: Optimizing Health Related Quality of Life Measurement in Adolescent and Young Adult Oncology: A Promising Solution (PROMIS AYA) - Aim 2
Brief Title: Optimizing Health Related Quality of Life Measurement in Adolescent and Young Adult Oncology
Status: Not yet recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00134827; R01CA218398 (NIH)
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Malignant Solid Neoplasm; Hematopoietic Neoplasms; Lymphatic System Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Participants will complete self-report questionnaires via Redcap. The questionnaires should take less than 30 minutes
  Interventions: Other: Surveys/Questionnaires

INTERVENTIONS:
Other: Surveys/Questionnaires — Participants will complete self-report questionnaires via Redcap. The questionnaires should take less than 30 minutes and will include the following options based on their relevance to each sample: 1) sociodemographic (including the comorbidity index) and clinical information, 2) newly developed item pools for body image, fertility, and financial burden, 3) legacy measures for body image, fertility, and financial burden, 4) the PROMIS AYA Health Status Profile, and 5) the PROMIS Global.

SUMMARY:
This study evaluates how adolescent and young adults with cancer in the U.S. and their loved ones respond to questions that will later be used with people who may have cancer and other chronic health conditions

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* To refine patient-reported outcome assessment tools of body image, fertility, and financial burden for PROMIS and evaluate assumptions for IRT consistent with PROMIS Scientific Standards (e.g., unidimensionality, local independence).
* To examine item-level properties to support computer adaptive testing and evaluate possible differential item functioning (DIF).

Secondary Objective

* To create short forms and examine convergent validity of the new body image, fertility, and financial burden short forms and item banks with corresponding legacy measures of those constructs.

OUTLINE: This is an observational study.

Participants complete surveys on study.

ELIGIBILITY:
AYAs with a cancer history (AYA-C)

Inclusion Criteria:

* Young adults between the ages of 15 to 39 years;
* First diagnosed with cancer during 15 to 39 years of age;
* Able to read and understand English;
* Live in the United States;
* Have a new cancer diagnosis and are receiving curative treatment OR are currently 0 to 10 years post-treatment.

Exclusion Criteria:

* Diagnosed with basal cell skin cancer; or
* Are currently receiving hospice care.

AYAs General Population (AYA-GP)

Inclusion Criteria:

* Young adults between the ages of 15 to 39 years;
* Able to read and understand English; and
* Live in the United States.

Caregivers of AYAs with cancer (AYA-Cg)

Inclusion Criteria:

* 18 years of age or older;
* Able to read and understand English;
* Live in the United States;
* Have a child/ward/partner for whom they have provided care, AND
* Their child/ward/partner is 15 to 25 years of age and meets the other eligibility criteria as an AYA participant with a cancer history (described above).

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adolescent young adults with and without cancer and caregivers of adolescent young adults with cancer.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Refining of Item Pools - Development of Four Item Banks | Up to study completion, up to approximately 2 years
  Upon completion of data analysis and study team review, investigators will have four unidimensional and locally independent, calibrated item banks: three for AYAs (body image, fertility, and financial burden) and one for caregivers (financial burden). In order to successfully calibrate an item bank, an n=500 is required per bank. In order to examine differential item functioning (DIF), a minimum n=200 per group is recommended. Our proposed sample sizes and specific subgroup accrual targets will be needed to calibrate multiple new item banks (body image, fertility, financial burden), evaluate DIF for various categories (age, gender, race, education) within our sample subgroups (AYAs with and without cancer), and to conduct confirmatory factor analysis (CFAs) on the item banks. In addition, the AYA sample the general population will serve as our reference to establish the mean and standard deviation for body image and fertility.

SECONDARY OUTCOMES:
Short Form Development Based on Item Bank Data | Up to study completion, up to approximately 2 years
  After the body image, fertility, and financial burden item banks have been calibrated from the primary outcome, short forms will be assembled by selecting the most informative (i.e., high measurement precision with little measurement error) and discriminating items (i.e., item response therapy (IRT) slopes that describe how well an item discriminates among individuals at different points along the measurement continuum) from each of the calibrated item banks. The convergent validity of the new PROMIS item banks and short forms will be examined using bivariate Pearson correlations with comparable constructs.

CONTACTS AND LOCATIONS:
Overall Officials: John Salsman, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No